CLINICAL TRIAL: NCT02243124
Title: A Study of Aezea® (Cenersen) in Transfusion Dependent Anemia Associated With Myelodysplastic Syndrome
Brief Title: A Study of Aezea® (Cenersen) in Transfusion Dependent Anemia Associated With Myelodysplastic Syndrome (MDS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Company went out of business
Sponsor: Eleos, Inc. (Industry)
Collaborators: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDS ELP9001
Record Dates: First submitted 2014-09-11; First posted 2014-09-17 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2017-01

CONDITIONS: Myelodysplastic Syndromes
Keywords: Anemia; Transfusion; AML; MDS; CLL; p53; erythropoiesis
MeSH Terms: conditions — Myelodysplastic Syndromes; Anemia | interventions — cenersen; OL(1)p53; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Active Comparator): cenersen IV infusion 0.3 mg/kg/day (0.1 mg/kg/h x 3 h x 4 days) for 6 cycles Administration of study drug will be over 4 consecutive days at the outset of each 28 day cycle for a total of 6 cycles for each patient. Dexamethasone 20 mg po weekly can be added after week 16 if stable disease but no Hematologic Improvement (HI) is observed.
  Interventions: Drug: cenersen; Drug: Dexamethasone
- Group 2 (Active Comparator): cenersen IV infusion 0.6 mg/kg/day (0.2 mg/kg/h x 3 h x 4 days) for 6 cycles Administration of study drug will be over 4 consecutive days at the outset of each 28 day cycle for a total of 6 cycles for each patient. Dexamethasone 20 mg po weekly can be added after week 16 if stable disease but no HI is observed.
  Interventions: Drug: cenersen; Drug: Dexamethasone
- Group 3 (Active Comparator): cenersen IV infusion 1.2 mg/kg/day (0.4 mg/kg/h x 3 h x 4 days) for 6 cycles Administration of study drug will be over 4 consecutive days at the outset of each 28 day cycle for a total of 6 cycles for each patient. Dexamethasone 20 mg po weekly can be added after week 16 if stable disease but no HI is observed.
  Interventions: Drug: cenersen; Drug: Dexamethasone

INTERVENTIONS:
Drug: cenersen — cenersen is a phosphorothioate antisense oligonucleotide that down-regulates the production of both wild-type and mutant p53, and has a RNase H-dependent mechanism of action
  Other Names: Ol(1)p53; EL625; Aezea
Drug: Dexamethasone — Optionally, Dexamethasone 20 mg po weekly can be added after week 16 if stable disease but no HI is observed.
  Other Names: Decadron; Maxidex; Ozurdex; Baycadron

SUMMARY:
The purpose of the study is to test the safety of six cycles of cenersen treatment and to begin to test the hypothesis that intermittent administration of cenersen may lead to a reduced dependence on transfusion.

DETAILED DESCRIPTION:
The study is a nonrandomized open-label treatment with varying doses of cenersen by intravenous administration to:

Primary

*To assess the safety profile and dose limiting toxicities (DLT) of cenersen for each of three increasing dose levels as stipulated by the protocol in patients with lower risk MDS defined as low or intermediate-1 risk by IPSS.

Secondary

* To determine the lowest pharmacologically active exposure from among three increasing dose levels as stipulated by the protocol that exhibits the desired activity on erythropoiesis after evaluation of all dose levels, and
* To determine if intermittent treatment with cenersen will reduce transfusion requirements for patients with lower risk MDS.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically or cytologically confirmed diagnosis of MDS according to WHO classification that meets IPSS low to intermediate-1 risk criteria.
* For patients with del(5q) MDS, documented del(5q) MDS by metaphase cytogenetics or FISH analysis with up to 1 additional cytogenetic abnormality other than 1 involving chromosome 7 or chromosome 17.
* Demonstrated refractoriness or intolerance to standard approved therapy (lenalidomide in del(5q) MDS patients & azanucleosides in non-del(5q)patients).
* Recovered from acute toxicities of other treatments (≤ Grade 2). All other MDS treatments discontinued at least 4 weeks prior to treatment except epoetin alpha (Procrit) 2 weeks.
* Ability to understand & willingness to sign a written informed consent document.
* Age ≥ 18 years at time of signing informed consent form.
* ECOG performance status ≤2.
* Life expectancy >4 weeks following initiation.
* Must meet following requirements:

  * total bilirubin: ≤2 x upper normal limit (UNL) (patients with Gilbert's disease are eligible, hyperbilirubinemia is intermittent & indirect)
  * AST(SGOT)/ALT(SGPT): ≤3 x UNL
  * creatinine: ≤2 x UNL
* <1% peripheral blood blasts.
* <10% bone marrow blasts.
* Medical history of RBC transfusion dependent anemia ≥4 units of RBCs during the 16 weeks prior to admin of study drug & ≥2 units of RBCs over prior 8 weeks (day -56 to day 1 prior to treatment; baseline period) for documented Hgb of ≤ 9g/dL (during baseline). Didn't have a 56 day RBC transfusion-free period during 16 weeks prior to administration of study drug.
* Teratogenic effects of cenersen are unknown, women of child-bearing potential & men must agree to use adequate contraception prior to study entry & for the duration of study participation.

Exclusion Criteria:

* Receiving MDS treatment except blood transfusion and/or iron chelation within 4 weeks prior to entering study or no recovery from adverse events due to agents administered more than 4 weeks earlier.
* no current or prior use of investigational agents within 4 weeks of study entry.
* Known history of malignancy diagnosed within 2 years other than non-melanoma skin cancer.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to cenersen.
* exclude use of acetaminophen or acetaminophen-containing medications from 1 day before to 1 day after completion of treatment. The active metabolite of acetaminophen, N-acetyl-p-benzoquinone imine (NAPQI), is known to block effects of cenersen & use of acetaminophen during treatment with study regimen has been associated with a failure to achieve a response in a past clinical trial of cenersen.
* Uncontrolled intercurrent illness that would limit compliance with study requirements.
* Pregnant women are excluded from this study. Breastfeeding should be discontinued if the mother is treated with cenersen
* HIV-positive patients on combination antiretroviral therapy are ineligible because of unknown potential for interactions with cenersen.
* Any condition, including presence of laboratory abnormalities, which places subject at unacceptable risk if s/he were to participate in study or confounds ability to interpret data from study according to investigator assessment.
* Therapy related MDS.
* Clinically significant anemia according to investigator's assessment due to factors such as iron, B12 or folate deficiencies, autoimmune or hereditary hemolysis or gastrointestinal bleeding.
* Received hematopoietic growth factors within specified limits prior to treatment (2 weeks for epoetin alpha (Procrit) & 4 weeks for darbepoetin alpha (Aranesp)).
* Active hepatitis B or C or other active liver disease.
* Chronic use (>2 weeks) of greater than physiologic doses of corticosteroid agent (dose equivalent to ≥10mg of prednisone) within 28 days of 1st day of study drug treatment & during treatment

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09-30 (Actual); Study Completion 2015-12-31 (Actual)

PRIMARY OUTCOMES:
1) Interventional Drug Safety: dose limiting toxicities (DLT) of cenersen for each of three increasing dose levels as stipulated by the protocol in patients with lower risk MDS defined as low or intermediate-1 risk by IPSS. | 6 months w/ 24 month follow-up
  Assessment of adverse events for each dosing level

SECONDARY OUTCOMES:
Reduction in RBC transfusions | 6 months w/ 24month follow-up
  Erythroid Response (HI-E) from the lowest pharmacologically active exposure after evaluation of all dose levels - Reduction in RBC transfusions by greater than or equal to 4 units/8 weeks triggered by a hemoglobin transfusion threshold lower than 9 g/dL when compared to the 8 week baseline for transfusion-dependent patients (where transfusion dependence is defined as 4 units or more RBCs in 8 weeks)
Improvement in Hemoglobin (Hb) levels | 6 months w/ 24 month follow-up
  Hematologic Improvement by Hb increase by ≥ 1.5 g/dL or more for at least 8 weeks and the patient is not transfusion-dependent.

CONTACTS AND LOCATIONS:
Overall Officials: Rami Komrokji, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

REFERENCES:
- [Background] Caceres G, McGraw K, Yip BH, Pellagatti A, Johnson J, Zhang L, Liu K, Zhang LM, Fulp WJ, Lee JH, Al Ali NH, Basiorka A, Smith LJ, Daugherty FJ, Littleton N, Wells RA, Sokol L, Wei S, Komrokji RS, Boultwood J, List AF. TP53 suppression promotes erythropoiesis in del(5q) MDS, suggesting a targeted therapeutic strategy in lenalidomide-resistant patients. Proc Natl Acad Sci U S A. 2013 Oct 1;110(40):16127-32. doi: 10.1073/pnas.1311055110. Epub 2013 Sep 16. PMID 24043769